CLINICAL TRIAL: NCT02257359
Title: A Phase 1, Open Label, Ascending Cohort, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Epelsiban and Its Metabolite in Healthy Female Volunteers Following Administration of Epelsiban
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Epelsiban in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201691
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Embryo Transfer
Keywords: Epelsiban; Healthy Female Volunteers; Safety; Tolerability; Oxytocin; Pharmacokinetics
MeSH Terms: interventions — epelsiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epelsiban Cohort 1 (Experimental): Subjects will receive 300 mg of epelsiban administered orally twice (every 12 hr) on Day 1 (total daily dose of 600 mg)
  Interventions: Drug: Epelsiban
- Epelsiban Cohort 2 (Experimental): Epelsiban dose for Cohort 2 will be determined based on data from Cohort 1, but will not exceed a total daily dose of 900 mg, administered orally in divided doses (450 mg every 12 hrs or 300 mg every 8 hrs).
  Interventions: Drug: Epelsiban
- Additional Cohorts TBD (to be decided) (Experimental): Subjects will be enrolled if determined necessary, based on data collected in Epelsiban Cohort 1 and Cohort 2
  Interventions: Drug: Epelsiban

INTERVENTIONS:
Drug: Epelsiban — Epelsiban will be supplied as a 25 mg white to off-white round direct compression oral tablet.

SUMMARY:
Epelsiban is a potent and selective oxytocin receptor antagonist in development for enhanced implantation rates during in-vitro fertilization (IVF). This study a non-randomized, open label study designed to assess the safety, tolerability and pharmacokinetics of additional repeat doses of epelsiban in healthy females, and will be the first dosing experience of greater than 200 milligram (mg) as a single dose with this compound. Data from this study will inform the selection of doses of epelsiban to be used in future clinical studies. This study will be composed of 3 periods: Screening, Treatment, and Follow-up. The total duration that a subject involved in the study will be up to 6 weeks. At least 2 cohorts of subjects will be enrolled in this study and cohorts will be conducted sequentially. Additional cohorts will be enrolled if determined necessary. A sufficient number of subjects will be screened for the study to obtain approximately 6 evaluable subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 55 years of age inclusive, at the time of consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, review of medications previously used, physical examination, laboratory tests and ECG.
* Body mass index (BMI) within the range 18-35 kilogram per square meter( kg/m^2) (inclusive).
* Female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential or postmenopausal.

Exclusion Criteria

* Alanine Transferase (ALT) and bilirubin >1.5x upper limit of normal(ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) > 450 milliseconds (msec). - History of regular alcohol consumption within 3 months of dosing on Day 1 defined as: an average weekly intake of >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of Study Treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2015-01-29 (Actual)

PRIMARY OUTCOMES:
Composite pharmacokinetic parameters of epelsiban and its metabolite (GSK2395448) | Up to Day 2
  Pharmacokinetic parameters including area under the plasma drug (and metabolite) concentration versus time curve (AUC[0-t], AUC[0- infinity], AUC[0-tau]), maximum observed concentration (Cmax), time to maximum observed plasma drug (and metabolite) concentration (tmax), and terminal half-life (t1/2), as data permit, will be analyzed. Blood samples for pharmacokinetic analysis will be collected on Day 1 (Morning pre-dose and 0.5hour(hr), 1 hr, 4 hr, 6hr, 8 hr, 12 hr post morning dose; evening pre-dose and 12.5 hr, 13 hr post morning dose) and Day 2 (16 hr and 24 hr post Day 1 morning dose).
Number of subjects with Adverse events (AEs) | Up to Day 12
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Assessment of clinical observations | Up to Day 12
Assessment of hematology parameters | Up to Day 12
  Hematology parameters include complete blood count with red blood cell indices, white blood cell count differential, hemoglobin, hematocrit and platelet count.
Assessment of clinical chemistry parameters | Up to Day 12
  Clinical chemistry parameters includes glucose, blood urea, creatinine, sodium, potassium, calcium, total protein, albumin, total bilirubin, direct bilirubin, alkaline phosphatase, alanine aminotransferase and aspartate aminotransferase.
Assessment of urinalysis by dipstick | Up to Day 12
  Urinalysis includes specific gravity, pH, glucose, protein, blood and ketones by dipstick. If blood or protein is abnormal microscopic examination will be done.
Assessment of vital sign measurements | Up to Day 12
  Vital sign measurements will include temperature, systolic and diastolic blood pressure and heart rate.
Assessment of 12-lead electrocardiogram (ECG) | Up to Day 12
  Triplicate 12-lead ECGs will be obtained at each timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Assessment of physical examination findings | Up to Day 12
  A physical examination will include, at a minimum, assessment of the cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight will also be measured

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mahar KM, Enslin MB, Gress A, Amrine-Madsen H, Cooper M. Single- and Multiple-Day Dosing Studies to Investigate High-Dose Pharmacokinetics of Epelsiban and Its Metabolite, GSK2395448, in Healthy Female Volunteers. Clin Pharmacol Drug Dev. 2018 Jan;7(1):33-43. doi: 10.1002/cpdd.363. Epub 2017 May 26. PMID 28556598
- See also: Results for study 201691 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201691?search=study&search_terms=201691#rs